CLINICAL TRIAL: NCT04935112
Title: A Phase 1 Study of the Effect of Acid-reducing Agents on the Pharmacokinetics of a Single Oral Dose of Sitravatinib in Healthy Adult Subjects
Brief Title: A Study to Explore the Effect of Acid-reducing Agents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 516-011
Record Dates: First submitted 2021-06-10; First posted 2021-06-22 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Healthy Adults
MeSH Terms: interventions — sitravatinib; Pantoprazole; Famotidine

STUDY DESIGN:
Intervention Model Description: 2 period crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 Treatment A (sitravatinib only) (Experimental): Period 1: A single oral dose of 100 mg sitravatinib on Day 1
  Interventions: Drug: Sitravatinib
- Group 1 Treatment B (sitravatinib and pantoprazole) (Experimental): Period 2: Oral pantoprazole once daily for 7 days (Days 1 to 7) and a single oral dose of 100 mg sitravatinib on Day 7
  Interventions: Drug: Sitravatinib; Drug: Pantoprazole
- Group 2 Treatment C (sitravatinib only) (Experimental): Period 1: A single oral dose of 100 mg sitravatinib on Day 1
  Interventions: Drug: Sitravatinib
- Group 2 Treatment D (sitravatinib and famotidine) (Experimental): Period 2: A single oral dose of 100 mg sitravatinib followed by a single oral dose of famotidine 40 mg approximately 2 hours after sitravatinib dose on Day 1
  Interventions: Drug: Sitravatinib; Drug: Famotidine

INTERVENTIONS:
Drug: Sitravatinib — 100 mg sitravatinib on Day 1
  Other Names: MGCD516
Drug: Pantoprazole — 40 mg QD on Day 1 to Day 7 of Period 2 in Group 1
  Other Names: Protonix
  Arms: Group 1 Treatment B (sitravatinib and pantoprazole)
Drug: Famotidine — 40 mg PO 2 hrs after sitravatinib in Period 2 of Group 2
  Other Names: Pepcid
  Arms: Group 2 Treatment D (sitravatinib and famotidine)

SUMMARY:
A Phase 1 Study of the Effect of Acid-reducing Agents on the Pharmacokinetics of a Single Oral Dose of Sitravatinib in Healthy Adult Subjects. The study is a single-center, open-label, 2-period, 2-treatment, fixed-sequence crossover, parallel-group study.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index between 18.0 and 32.0 kg/m2, inclusive.
* In good health, determined by no clinically significant findings from medical history, physical examination, 12 lead ECG, vital sign measurements, and clinical laboratory evaluations at screening and/or check-in, as assessed by the investigator (or qualified designee).
* Females of childbearing potential will not be pregnant or lactating and must have a negative result on an approved pregnancy test at screening and check-in. Females of childbearing potential must agree to use contraception.
* Male subjects must agree to use contraception.
* Able to comprehend and willing to sign an ICF and to abide by the study restrictions.

Key Exclusion Criteria:

* Significant history of clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator.
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, any components of the IMP, or other substance (not including seasonal allergies), unless approved by the investigator.
* History of intestinal disease, inflammatory bowel disease, major gastric surgery, or other gastrointestinal conditions (eg, uncontrolled nausea, vomiting, malabsorption syndrome) likely to alter absorption of study treatment or result in inability to swallow oral medications. (Uncomplicated appendectomy and hernia repair are allowed. Cholecystectomy is not allowed.)
* History of Gilbert's syndrome or suspicion of Gilbert's syndrome based on elevated total and indirect bilirubin (may be confirmed by repeat).
* Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to study drug administration on Day 1 of Period 1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - Cmax (sitravatinib) | Up to Day 7 after dosing
  Maximum observed plasma concentration
Pharmacokinetics - AUC∞ (sitravatinib) | Up to 72 hours after dosing
  Area under the plasma concentration-time curve from time zero extrapolated to infinity
Pharmacokinetics - AUClast (sitravatinib) | Up to 72 hours after dosing
  Area under the curve from time zero to the last measured time point

SECONDARY OUTCOMES:
Adverse Events (AEs) | Up to 9 weeks from screening
  Incidence and severity of AEs

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Chin, MD, Study Director — Mirati Therapeutics Inc.
Locations (1):
- Covance Clinical Research Unit Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No